CLINICAL TRIAL: NCT01431482
Title: Evaluation of the Composition of Human Milk and Health Outcomes in Children
Status: Completed | Type: Observational
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: 6010
Record Dates: First submitted 2011-06-07; First posted 2011-09-09 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2013-05

CONDITIONS: Respiratory Symptoms; Signs and Symptoms, Digestive; Anemia
Keywords: skin symptoms
MeSH Terms: conditions — Signs and Symptoms, Respiratory; Signs and Symptoms, Digestive; Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human milk samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is an evaluation of the composition of human milk and health outcomes in children.

ELIGIBILITY:
Inclusion Criteria:

* Human milk samples from mothers from a larger birth co-hort study
* Health outcomes of children from mothers from a larger birth co-hort study from birth through two years of age

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children up to 2 years of age
Sampling Method: Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Incidence of infectious and allergic Gastrointestinal events through 2 years of age | 2 years of age
  Number of incidences of infectious and allergic Gastrointestinal events for each participant through 2 years of age

SECONDARY OUTCOMES:
Incidence of infectious and allergic respiratory events through 2 years of age | 2 years of age
  Number of incidences of infectious and allergic respiratory events for each participant through 2 years of age
anthropometric measurements | 2 years of age
  participants' weight, length and head circumference
Incidence of anemia in first 2 years of age | 2 years of age
  Hemoglobulin measurement

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Ribeiro, Jr, M.D., Principal Investigator — Federal University of Bahia School of Nutrition